CLINICAL TRIAL: NCT00129701
Title: Proposal to Study Whether we Can Reduce Hospital Attendance by Those With Respiratory Conditions Without Compromising Care by the Use of Telephone Consultation
Brief Title: Can we Reduce Hospital Attendance Without Compromising Care by the Use of Telephone Consultation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NHLICX3510
Record Dates: First submitted 2005-08-11; First posted 2005-08-12 (Estimated); Results first posted 2020-01-23 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Asthma; COPD; Sleep Apnea Syndromes; Interstitial Lung Diseases; Bronchiectasis
Keywords: phone consultation in secondary care
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive; Sleep Apnea Syndromes; Lung Diseases, Interstitial; Bronchiectasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients attending (Experimental): Patients recruited to have a telephone consultation and then at the next appointment a face-to-face appointment
  Interventions: Procedure: Telephone consultation

INTERVENTIONS:
Procedure: Telephone consultation

SUMMARY:
Consultation time in busy respiratory clinics is inevitably limited and attendance is often disruptive to patients' lives; involves time, expense, travel, and waiting; and can have effects upon occupation. Published work suggests that patient satisfaction with telephone consultations is high and this subject has recently been extensively reviewed by one of the study investigators. In respiratory medicine there is United States (US) data to suggest that the regular telephoning of adolescents with asthma by a specialist nurse can reduce unscheduled use of health service resources. In the United Kingdom (UK), a randomised, controlled trial in primary care has shown that, compared to face to face consultations, use of the telephone can enable greater numbers of patients with asthma to be reviewed. Another of the study investigators has undertaken a feasibility study in a general respiratory clinic and has shown the concept of alternating face to face consultation with telephone consultation to be acceptable to over 80% of patients. Over one third were assessed to be suitable in that they did not need to attend the clinic for either physical examination or for investigations. It is therefore proposed to evaluate the feasibility, acceptability, time savings and safety of the use of telephone consultation in 3 respiratory clinics in the Department of Respiratory Medicine at Charing Cross Hospital.

DETAILED DESCRIPTION:
Patients to be included in the study would be those attending 3 respiratory clinics. The patients would be asked if they were willing to have a telephone consultation instead of their next face to face consultation and this would be explained to them.

"Many patients attending a Chest Clinic need to do so only once. For others their condition merits regular review. Most of these people need to come to the clinic because they need chest x-rays, blood tests or breathing tests. However some patients return for review of their condition without needing any specialist investigations. We are keen to assess what proportion of our patients would be suitable for telephone consultations rather than face to face consultations and to see what advantages there might be for both patients and doctors. We are therefore interested to assess the use of telephone consultation where suitable and would like to know if you would be willing to try telephone consultation for your next appointment. In the case of telephone consultation you would be offered a day, date and time at which you would be phoned. Your consultant, would then ring you him or herself within half an hour of the appointed time {and procedurally it has been agreed by the trial participants that if, for any reason, during the trial period they are delayed with the previous patient they will excuse themselves to telephone the following patient to say that they have been delayed and they will ring them back within 15 minutes, for example} and with your clinical notes in front of them he or she would enquire in the usual way regarding how you feel, ask about your symptoms and give advice regarding any concerns you may have or advise regarding changes in treatment. You would subsequently receive a copy of the letter summarising the telephone consultation when it was sent to your general practitioner. If the telephone consultation suggested that you needed to be seen in the clinic you would be offered an appointment within two weeks of the telephone call."

Demographic details and disease diagnosis would be recorded, for those not deemed suitable or for those not wishing to take part and they would continue to attend traditional face to face consultations. Those having a telephone consultation would subsequently revert to traditional consultation pending results of the trial. Frequency of planned consultation would be as per the consultant's usual practice.

Procedurally, it was agreed that for those patients agreeing to have their next consultation by telephone, the doctor would check the phone number which they wished for the investigators to use and this would be inserted in the notes at the end of the previous consultation with a large black box around it, so that it could easily be spotted at the time of the telephone consultation.

For all patients the following observations would be made: length of the telephone consultation, fail to be available when telephoned rate, and length of each face to face consultation.

For each face to face consultation the following information would be recorded: the time they left home; time of arrival at hospital, time spent waiting for consultation, expense of attendance, both travel costs but also any indirect costs such as babysitting charges and loss of earnings. For each telephone consultation the number of patients having to be reviewed within the next 2 weeks of the telephone consultation would be recorded, whether such expedited follow up was at the patient's or the doctor's behest.

After both the telephone consultation and their subsequent face to face consultation the patients would be asked to complete the post consultation patient satisfaction questionnaire, the MISS 21 questionnaire and the Howie Enablement Instrument. Patients would be posted these scales by first class post on the day of a telephone consultation and handed them for completion after a face to face consultation and on each occasion they would be given a stamped addressed envelope in which to return the completed scores.

ELIGIBILITY:
Inclusion Criteria:

Patients who had already attended a respiratory clinic on at least two occasions and in whom it was perceived that there was a need for continued follow up in a hospital clinic with review needed more often than once per year Patients with no need for physical examinations or investigations such as chest X-rays, blood tests or lung function tests at every attendance Patients who had access to a confidential telephone line Patients who had no mental, hearing or linguistic problems

Exclusion criteria

New patients or those who need frequent follow up Patients with mental or cognitive issues Patients requiring physical examination and testing.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2003-11 (Actual); Primary Completion 2005-10 (Actual); Study Completion 2006-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martyn R Partridge, MD FRCP, Principal Investigator — NHLI Imperial College
Locations (1):
- NHLI Imperial College, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pal B. Following up outpatients by telephone: pilot study. BMJ. 1998 May 30;316(7145):1647. doi: 10.1136/bmj.316.7145.1647. No abstract available. PMID 9603747
- [Background] Car J, Sheikh A. Telephone consultations. BMJ. 2003 May 3;326(7396):966-9. doi: 10.1136/bmj.326.7396.966. No abstract available. PMID 12727771
- [Background] Greineder DK, Loane KC, Parks P. Reduction in resource utilization by an asthma outreach program. Arch Pediatr Adolesc Med. 1995 Apr;149(4):415-20. doi: 10.1001/archpedi.1995.02170160069010. PMID 7704170
- [Background] Pinnock H, Bawden R, Proctor S, Wolfe S, Scullion J, Price D, Sheikh A. Accessibility, acceptability, and effectiveness in primary care of routine telephone review of asthma: pragmatic, randomised controlled trial. BMJ. 2003 Mar 1;326(7387):477-9. doi: 10.1136/bmj.326.7387.477. PMID 12609944
- [Background] Partridge MR. An assessment of the feasibility of telephone and email consultation in a chest clinic. Patient Educ Couns. 2004 Jul;54(1):11-3. doi: 10.1016/S0738-3991(03)00166-6. PMID 15210254
- [Result] Roberts NJ, Partridge MR. Telephone consultations in secondary care. Respir Med. 2007 Aug;101(8):1665-9. doi: 10.1016/j.rmed.2007.03.003. Epub 2007 Apr 19. PMID 17448649

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients Attending: Patients recruited to have a telephone consultation and then at the next appointment a face-to-face appointment
  Telephone consultation
Period: Overall Study
Arm/Group | Patients Attending
Started | 104
Completed | 71
Not Completed | 33
Not completed — Withdrawal by Subject | 33

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were not collected
Arm/Group | Patients Attending
Number analyzed (Participants) | 0
Age, Customized
Sex/Gender, Customized
Race and Ethnicity Not Collected — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Patient Satisfaction
Description: MISS-21 satisfaction scale, The 21 items are scored using a 7-point Likert scale with responses ranging from 1 ("Very strongly disagree") to 7 ("Very strongly agree"). Maximum is 147 Very strong satisfaction - best outcome, minimum 21 very strong dissatisfaction.
Time Frame: After consultation within 1 months
Population: Participants who attended both types of consultations
Measure: Mean (Standard Deviation); unit: score on scale
Groups:
- Telephone Consultation: Participants attended to a Telephone consultation
- Face-to-face Consultation: Participants attended to a Face-to-face consultation
Arm/Group | Telephone Consultation | Face-to-face Consultation
Number analyzed (Participants) | 45 | 45
score on scale | 114.3 (14) | 116.8 (15)
Statistical Analysis 1: Comparison: Telephone Consultation vs Face-to-face Consultation; Test type: Superiority; p = 0.064, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Patients Needing Expedited Follow up
Description: Number of participants who were telephoned and needed expedited follow-up
Time Frame: After phone consultation within 2 weeks
Population: Number of participants who were telephoned at the pre-arranged time and they were available
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Attending
Number analyzed (Participants) | 71
Participants | 4

3. Primary Outcome: Costs Associated With Traditional Face to Face Consultation
Description: Patient costs attending hospital appointments compare to phone consultations
Time Frame: 1 year
Population: No data collected
Arm/Group | Patients Attending
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Patients Attending
All-Cause Mortality (participants affected / at risk) | 0/104
Serious Adverse Events (participants affected / at risk) | 0/104
Other Adverse Events (participants affected / at risk) | 0/104

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes